CLINICAL TRIAL: NCT01979913
Title: An Open, Non-randomized Pilot Study on the Effect of Preservative Free Tafluprost (Saflutan® Augentropfen) in Patients With Ocular Hypertension or Primary Open Angle Glaucoma With an Uncontrolled Intraocular Pressure of 30 mmHg and More
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Anton Hommer (Other)
Responsible Party: Sponsor-Investigator, Dr. Anton Hommer, Dr. med. univ., Ordination Dr. Hommer
Organization: Ordination Dr. Hommer (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPHT-260213
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Primary Open Angle Glaucoma; Ocular Hypertension; Tafluprost; Saflutan; Intraocular pressure; Preservative free; Single dose unit
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — tafluprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with POAG or OHT (Experimental): Patients with primary open angle glaucoma or ocular hypertension
  Interventions: Drug: Saflutan® 15 microgram/ml Augentropfen im Einzeldosisbehältnis

INTERVENTIONS:
Drug: Saflutan® 15 microgram/ml Augentropfen im Einzeldosisbehältnis
  Other Names: Tafluprost

SUMMARY:
Increased intraocular pressure (IOP) has been identified as the most important risk factor for the development and the progression of glaucoma. Data from large interventional studies have shown that a decrease of IOP is associated with a reduced risk of progression of the disease. This underlines the importance of a potent and save IOP lowering therapy. The introduction of preservative free tafluprost offers a new treatment possibility using a potent topical prostaglandin analogue without the disadvantages of a co-administered preservative. The current study seeks to investigate the effect of an 8 week therapy with preservative free tafluprost on intraocular pressure in patients with ocular hypertension or primary open angle glaucoma having an IOP of 30 mmHg or more.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Diagnosed primary open angle glaucoma and an IOP of 30mmHg or more in at least 1 eye at visit 1 at 8 am
* Patients with ocular hypertension as defined as an IOP of 30mmHg or more and normal findings in the visual field and the optic nerve head

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks before the screening visit
* Severe visual field loss as defined as an MD of -15 or worse
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition that will interfere with the study aim as judged by the clinical investigator
* Presence or history of a severe ocular condition that will interfere with the study aim as judged by the clinical investigator
* Wearing of contact lenses
* Topical treatment with any ophthalmic drug in the 4 weeks preceding the study except glaucoma medication or topical lubricants
* Ocular infection
* Ocular surgery in the 6 months preceding the study
* Pregnancy, planned pregnancy or lactating
* Contraindication against the use of topical prostaglandin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 8 weeks
  Intraocular pressure will be measured at baseline, after 4 weeks and after 8 weeks at 8:00 am and 6:00 pm on each study day

CONTACTS AND LOCATIONS:
Locations (1):
- Ordination Dr. Hommer, Vienna, Vienna, Austria